CLINICAL TRIAL: NCT06572319
Title: Phase I/II Clinical Study of the Combination of Disitamab Vedotin and Trastuzumab in the Treatment of HER2 Positive Gastric/Gastroesophageal Junction Tumors With Previous Systemic Therapy Failure
Brief Title: Disitamab Vedotin Plus Trastuzumab in Patients With HER2 Positive GC/GEJ Patiens
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-278
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: HER2-positive Gastric Cancer; HER2-positive Gastroesophageal Junction Adenocarcinoma
Keywords: HER-2; ADC; Disitamab Vedotin; trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ⅰ/Ⅱ： Disitamab Vedotin(RC48) Plus Tratuzumab (Experimental): Dose exploration： Disitamab Vedotin（RC48）: 2.5mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle.
  Tratuzumab:"3+3"Design，1mg/kg Q2W，2.5mg/kg Q2W，4mg/kg Q2W Dose expansion： Disitamab Vedotin（RC48）: 2.5mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle.
  Tratuzumab: RP2D
  Interventions: Drug: Disitamab Vedotin(RC48) Plus Tratuzumab

INTERVENTIONS:
Drug: Disitamab Vedotin(RC48) Plus Tratuzumab — Disitamab Vedotin: 2.5mg/kg，ivgtt，D1, every 2 weeks for a treatment cycle. Tratuzumab: RP2D，ivgtt，D1, every 2 weeks for a treatment cycle.

SUMMARY:
This trial is a single center, single arm, open label clinical study aimed at evaluating the efficacy and safety of the combination therapy of Disitamab Vedotin and trastuzumab in the treatment of advanced HER-2 positive gastric/gastroesophageal junction tumors

DETAILED DESCRIPTION:
In a specific tumor area, the absorption of antibodies is driven by its blood vessels or permeable surface, while the microscopic distribution depends on the number of binding sites available for the specific antibody. Due to the much faster binding rate of antibodies to their targets than their diffusion rate, their penetration into tumor tissue is severely limited (such as binding site barriers). This will limit the drug's penetration into the tumor before the antibody reaches saturation dose. Due to the toxicity brought by the toxins carried by ADC itself (toxin shedding, non-specific endocytosis, or on target, off tumor toxicity), its dose will be relatively reduced compared to naked antibodies. By adding naked antibodies or directly reducing DAR, the dose of ADC can be increased to overcome the binding site barrier and improve the tumor penetration of antibody drugs. In theory, if the antibody dose is large enough, the antibody will reach all (accessible) binding points within the tumor and saturate both the interior and periphery of the tumor.

In addition, in addition to ADC drugs, chemotherapy, immunotherapy, targeted therapy, and other options are also available for HER2 positive gastric cancer posterior line, but the efficacy is still unclear. Therefore, it is urgent to explore new treatment options to further improve the efficacy of this special population.

Therefore, we designed this Phase I/II clinical trial to explore whether the combination of RC48 and naked anti trastuzumab currently on the market can improve efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form; 2.18-75 years old (including 18 years old, excluding 75 years old), gender not limited; 3. The pathological histology confirmed by pathology is adenocarcinoma of the gastric/gastroesophageal junction; 4. HER2 positive tumor criteria (primary tumor or metastatic lesion, HER2 positive is defined as IHC 2+/FISH+(HER2: CEP17 ratio ≥ 2.0) or IHC (3+). Using the criteria for interpreting HER2 in gastric cancer 5. Recurrent or metastatic diseases that cannot be surgically treated, with at least one measurable lesion (RECIST 1.1 criteria) in the subject and an estimated survival time of at least 12 weeks; 6. ECOG score ranges from 0 to 1 points; 7. At least first-line systemic therapy has failed (regardless of whether it includes anti-HER2 monoclonal antibody therapy); 8. Having sufficient bone marrow, liver and kidney function:

* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 90 × 109/L, or
* hemoglobin ≥ 9g/dL;
* ALT or AST levels without liver metastasis are less than 2.5 times the upper limit of the normal range; When liver metastasis occurs, ALT or AST is less than 5 times the upper limit of the normal range; Serum bilirubin is 1.5 times lower than the upper limit of the normal reference range;
* Serum creatinine is lower than 1.5 times the upper limit of the normal reference range or creatinine clearance rate is ≥ 40ml/min; 9. Women of childbearing age and their spouses are willing to use effective contraceptive methods within the last 7 months of treatment.

Exclusion Criteria:

1. Known to be allergic to the received therapeutic drugs or excipients;
2. Baseline LVEF<50% (measured by echocardiography or MUGA);
3. Previously received treatment with anti-HER2 ADC drugs;
4. Individuals who have undergone systemic immunotherapy, biologic therapy, or participated in any clinical drug trials within the past 2 weeks;
5. Those who have undergone surgery within 3 weeks before the start of the experimental treatment and have not fully recovered;
6. Patients with uncontrolled central nervous system (CNS) metastases or epilepsy requiring medication treatment;
7. Serious systemic diseases. Such as infected or uncontrolled diabetes;
8. Suffering from other malignant tumors within 5 years, except for non melanoma skin cancer and cervical carcinoma in situ;
9. Clinically symptomatic active coronary heart disease, cardiomyopathy, or congestive heart failure, NYHA III-IV; uncontrolled hypertension (systolic blood pressure>180 mmHg or diastolic blood pressure>100 mmHg), clinically symptomatic heart valve disease, or high-risk arrhythmia;
10. Patients receiving long-term or high-dose corticosteroid treatment (inhaled steroids or short-term oral steroids are allowed to resist vomiting or promote appetite)
11. Individuals without legal capacity, those whose medical or ethical reasons affect the continuation of research;
12. Pregnant and lactating female patients, or those who wish to become pregnant during treatment;
13. Uncontrolled pleural and peritoneal effusion;
14. There is a persistent infection of>level 2 (CTC-AE 4.0); Wounds, ulcers, or fractures that cannot heal, or patients with a history of organ transplantation;
15. There are unresolved toxicity levels>1 caused by any previous treatment/procedure (CTC-AE 4.0, excluding hair loss, anemia, and hypothyroidism);
16. After comprehensive assessment of the patient's condition by the researchers, it is deemed that they are not suitable to participate in this study;
17. Simultaneously participating in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 12 months
  he number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)
Progression-free survival (PFS) | up to 12 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Disease control rate (DCR) | up to 12 months
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Incidence of Treatment-Emergent 3/4 Adverse Events | up to 12 months after enrollment or study close
  Number and percentage of participants with Adverse Events (any Grade and Grade 3/4)

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No